CLINICAL TRIAL: NCT00281593
Title: A Randomized, Double-blind, Double-dummy, Placebo-controlled, 3x4 Factorial Design Trial to Evaluate Telmisartan 20 and 80 mg Tablets in Combination With Ramipril 1.25, 10, and 20 mg Capsules After Eight Weeks of Treatment in Patients With Stage I or II Hypertension, With an ABPM Sub-study
Brief Title: Telmisartan (Micardis) and Ramipril (Altace) - Factorial Design Study for the Treatment of Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Purpose: Treatment
Other Study IDs: 1236.1
Record Dates: First submitted 2006-01-24; First posted 2006-01-25 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan; Ramipril

INTERVENTIONS:
Drug: Telmisartan
Drug: Ramipril

SUMMARY:
To identify dose combinations of telmisartan and ramipril that are more effective in reducing diastolic blood pressure than each of the respective monotherapies in patients with Stage I or II hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients >=18 years of age with Stage I or II hypertension defined as:
* a mean seated cuff diastolic blood pressure >=95 and <=119 mmHg Main

Exclusion Criteria:

* Pregnant
* breast-feeding
* unwilling to use birth control during the study
* secondary hypertension
* SBP>=180 mmHg
* DBP>=120 mmHg
* severe renal dysfunction
* hepatic insufficiency
* stroke within the last 6 months
* myocardial infarction, cardiac surgery, percutaneous transluminal coronary angioplasty, unstable angina or coronary artery bypass graft within the past three months
* unstable or uncontrolled diabetes
* history of angioedema of either of the study drugs, and hypersensitivity to the study drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1354 (Actual)
Dates: Start 2006-04; Primary Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in seated trough Diastolic Blood pressure after 8 weeks of treatment

SECONDARY OUTCOMES:
Change from baseline in systolic blood pressure after 8 weeks of treatment Percentage of patients responding to treatment Changes from baseline in diastolic and systolic blood pressure hourly means over the 24 hour dosing interval as measured by ABPM

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (119):
- United States (70):
  - 1236.1.511 Boehringer Ingelheim Investigational Site, Glendale, Arizona
  - 1236.1.574 Boehringer Ingelheim Investigational Site, Tempe, Arizona
  - 1236.1.501 Boehringer Ingelheim Investigational Site, Tucson, Arizona
  - 1236.1.557 Boehringer Ingelheim Investigational Site, Tucson, Arizona
  - 1236.1.523 Boehringer Ingelheim Investigational Site, Buena Park, California
  - 1236.1.514 Boehringer Ingelheim Investigational Site, Concord, California
  - 1236.1.560 Boehringer Ingelheim Investigational Site, Encinitas, California
  - 1236.1.573 Boehringer Ingelheim Investigational Site, Long Beach, California
  - 1236.1.516 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1236.1.529 Boehringer Ingelheim Investigational Site, Roseville, California
  - 1236.1.519 Boehringer Ingelheim Investigational Site, Tustin, California
  - 1236.1.543 Boehringer Ingelheim Investigational Site, Westlake Village, California
  - 1236.1.528 Boehringer Ingelheim Investigational Site, Boulder, Colorado
  - 1236.1.530 Boehringer Ingelheim Investigational Site, Farmington, Connecticut
  - 1236.1.572 Boehringer Ingelheim Investigational Site, DeLand, Florida
  - 1236.1.577 Boehringer Ingelheim Investigational Site, Hialeah, Florida
  - 1236.1.526 Boehringer Ingelheim Investigational Site, Jupiter, Florida
  - 1236.1.527 Boehringer Ingelheim Investigational Site, Largo, Florida
  - 1236.1.503 Anchor Research Center, Naples, Florida
  - 1236.1.520 Boehringer Ingelheim Investigational Site, New Port Richey, Florida
  - 1236.1.571 Boehringer Ingelheim Investigational Site, Pembroke Pines, Florida
  - 1236.1.565 Boehringer Ingelheim Investigational Site, Blue Ridge, Georgia
  - 1236.1.538 Boehringer Ingelheim Investigational Site, Meridian, Idaho
  - 1236.1.532 Boehringer Ingelheim Investigational Site, Peoria, Illinois
  - 1236.1.553 Boehringer Ingelheim Investigational Site, Avon, Indiana
  - 1236.1.546 River Cities Cardiology Research Inst of Middle America, Jeffersonville, Indiana
  - 1236.1.563 Boehringer Ingelheim Investigational Site, Valparaiso, Indiana
  - 1236.1.517 Boehringer Ingelheim Investigational Site, Newton, Kansas
  - 1236.1.531 Boehringer Ingelheim Investigational Site, Wichita, Kansas
  - 1236.1.566 Boehringer Ingelheim Investigational Site, Richmond, Kentucky
  - 1236.1.551 Boehringer Ingelheim Investigational Site, Auburn, Maine
  - 1236.1.536 Boehringer Ingelheim Investigational Site, Haverhill, Massachusetts
  - 1236.1.576 Boehringer Ingelheim Investigational Site, North Dartmouth, Massachusetts
  - 1236.1.561 Clinical Research Center of Cape Cod, West Yarmouth, Massachusetts
  - 1236.1.555 Boehringer Ingelheim Investigational Site, Cadillac, Michigan
  - 1236.1.509 Boehringer Ingelheim Investigational Site, Troy, Michigan
  - 1236.1.541 Boehringer Ingelheim Investigational Site, Excelsior Springs, Missouri
  - 1236.1.556 Boehringer Ingelheim Investigational Site, Las Vegas, Nevada
  - 1236.1.525 Physicians Research Center, LLC, Toms River, Toms River, New Jersey
  - 1236.1.508 Boehringer Ingelheim Investigational Site, Albuquerque, New Mexico
  - 1236.1.522 Boehringer Ingelheim Investigational Site, Albuquerque, New Mexico
  - 1236.1.542 Boehringer Ingelheim Investigational Site, Albuquerque, New Mexico
  - 1236.1.547 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 1236.1.567 Boehringer Ingelheim Investigational Site, Columbus, Ohio
  - 1236.1.515 Boehringer Ingelheim Investigational Site, Kettering, Ohio
  - 1236.1.575 Boehringer Ingelheim Investigational Site, Tulsa, Oklahoma
  - 1236.1.554 Boehringer Ingelheim Investigational Site, Corvallis, Oregon
  - 1236.1.524 Boehringer Ingelheim Investigational Site, Eugene, Oregon
  - 1236.1.544 Boehringer Ingelheim Investigational Site, Medford, Oregon
  - 1236.1.545 Boehringer Ingelheim Investigational Site, Portland, Oregon
  - 1236.1.569 Boehringer Ingelheim Investigational Site, Erie, Pennsylvania
  - 1236.1.505 Ledeeach Family Medicine, Harleysville, Pennsylvania
  - 1236.1.564 Boehringer Ingelheim Investigational Site, Tipton, Pennsylvania
  - 1236.1.534 Boehringer Ingelheim Investigational Site, Cumberland, Rhode Island
  - 1236.1.539 Boehringer Ingelheim Investigational Site, Spartanburg, South Carolina
  - 1236.1.568 Boehringer Ingelheim Investigational Site, Carrollton, Texas
  - 1236.1.549 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1236.1.559 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1236.1.548 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 1236.1.550 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 1236.1.570 Boehringer Ingelheim Investigational Site, The Colony, Texas
  - 1236.1.510 Boehringer Ingelheim Investigational Site, Salt Lake City, Utah
  - 1236.1.513 Boehringer Ingelheim Investigational Site, Salt Lake City, Utah
  - 1236.1.521 Boehringer Ingelheim Investigational Site, Salt Lake City, Utah
  - 1236.1.512 Boehringer Ingelheim Investigational Site, Sandy City, Utah
  - 1236.1.535 Boehringer Ingelheim Investigational Site, Sandy City, Utah
  - 1236.1.502 Boehringer Ingelheim Investigational Site, Falls Church, Virginia
  - 1236.1.504 Boehringer Ingelheim Investigational Site, Madison, Wisconsin
  - 1236.1.540 Boehringer Ingelheim Investigational Site, Madison, Wisconsin
  - 1236.1.562 Boehringer Ingelheim Investigational Site, Menomonee Falls, Wisconsin
- Argentina (21):
  - 1236.1.601 Boehringer Ingelheim Investigational Site, Buenos Aires
  - 1236.1.604 Boehringer Ingelheim Investigational Site, Buenos Aires
  - 1236.1.605 Boehringer Ingelheim Investigational Site, Buenos Aires
  - 1236.1.610, Buenos Aires
  - 1236.1.612, Buenos Aires
  - 1236.1.619, Capital Federal,Buenos Aires
  - 1236.1.608, Capital Federal
  - 1236.1.618 Hospital Ramos Mejia, Capital Federal
  - 1236.1.615, CordobaCordoba
  - 1236.1.611, Corrientes
  - 1236.1.603 Boehringer Ingelheim Investigational Site, Córdoba
  - 1236.1.606, Córdoba
  - 1236.1.613, Córdoba
  - 1236.1.614, Córdoba
  - 1236.1.624 Instituto de Investigaciones Clínicas, Mar del Plata
  - 1236.1.609, Presidente Derqui
  - 1236.1.620 DIM - Clinica Privada, Ramos Mejía
  - 1236.1.622 Hospital San Bernardo, Salta
  - 1236.1.621 Clinica del Torax y Especialidades, Santa Fe
  - 1236.1.602 Boehringer Ingelheim Investigational Site, Villa Carlos Paz
  - 1236.1.616, Zárate
- Canada (11):
  - 1236.1.202 North Road Medical Centre, Coquitlam, British Columbia
  - 1236.1.208 Shoppers Drug Mart Building, Bay Roberts, Newfoundland and Labrador
  - 1236.1.206 77 Commonwealth Avenue, Mount Pearl, Newfoundland and Labrador
  - 1236.1.215 Cowan Avenue Medical Clinic, St. John's, Newfoundland and Labrador
  - 1236.1.203 MSHJ Research Associates, Halifax, Nova Scotia
  - 1236.1.210 Hamilton Medical Research, Hamilton, Ontario
  - 1236.1.204 Dr. Ivan Jagas, Kitchener, Ontario
  - 1236.1.209 St. Joseph Cardiovascular Inc, Ottawa, Ontario
  - 1236.1.207 Dr. Michael O'Mahony, Sarnia, Ontario
  - 1236.1.205 Ctr. Hospital U Quebec- Pav CHUL, Sainte-Foy, Quebec
  - 1236.1.211 Royal University Hospital, Saskatoon, Saskatchewan
- Chile (2):
  - 1236.1.106 Hospital Dr. Sótero del Río, Puente Alto, Santiago de Chile
  - 1236.1.103 Oficina 312 E (Cardiology Division), Santiago
- Mexico (10):
  - 1236.1.301 Fracc. Magallanes, Acapulco Guerrero
  - 1236.1.304 Fracc Agricultura, Aguascalientes
  - 1236.1.311 Hospital de Especialidades Miguel Hidalgo, Aguascalientes
  - 1236.1.305 Especialidades Médicas del sol, Col Ciudad de Sol Zapopan
  - 1236.1.310 Departamento de Hemodinamia, Col. Magdalena de Las Salinas
  - 1236.1.307 Consultorio: Aurelio L, Guadalajara
  - 1236.1.306, México D.F
  - 1236.1.308 Hospital Central "Dr. Ignacio Morones Prieto", San Luis Potosí City
  - 1236.1.302, Torreón
  - 1236.1.303, Veracruz
- Peru (5):
  - 1236.1.401 Unidad de Investigacion, Bella Vista, Callao,
  - 1236.1.405, San Borja
  - 1236.1.402, San Isidro
  - 1236.1.403, San Isidro
  - 1236.1.404, San Isidro

REFERENCES:
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/22272064